CLINICAL TRIAL: NCT03849235
Title: A Pathophysiological Study of the Postprandial Human Liver (PLS)
Acronym: PLS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Lise Gluud, Consultant hepatologist, Copenhagen University Hospital, Hvidovre
Other Study IDs: H-18052725
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Cirrhosis; Fatty Liver
MeSH Terms: conditions — Fibrosis; Fatty Liver | interventions — Glucagon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood tests and liver tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Standardised meal or glucagon — Standardised meal (Nutridrink, Nutricia, 300 kcal, 18.4 g carbohydrates, 5.8 g fat, 12 g protein) or 1mg glucagon

SUMMARY:
Fatty liver disease is a globally widespread disease The identification of valid biomarkers and targets for potential treatments requires in-depth knowledge about the pathophysiology of the postprandial liver. The study will consist of five work packages (WP) including blood tests and liver biopsies taken after fasting or ingestion of a standardized meal in: healthy controls (WP 1), patients with NAFLD (WP 2), and patients with cirrhosis (WP 3) ; before and after a standardised meal in healthy controls (WP 4), and before and after glucagon in healthy controls (WP5)

ELIGIBILITY:
Healthy participants (WP 1 , WP 4 , WP 5 )

Inclusion criteria: Healthy adults, 20 - 40 years old, non-smoker, BMI 20-25 kg/m2 , no chronical illnesses, no medication.

Exclusion criteria: Blood donation within the past 3 months, acute illness within 2 weeks

NAFLD ( WP 2)

Inclusion criteria: Patients with clinical diagnosis of NAFL and indication for liver biopsy Exclusion criteria: Malignant disease, acute illness within the past 2 weeks.

Cirrhosis (WP 3)

Inclusion criteria: Patients with clinical diagnosis of cirrhosis and indication for liver biopsy.

Exclusion criteria:Malignant disease, acute illness within the past 2 weeks.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will include partcipants with suspected NAFLD or cirrhosis based on clinical assessments referred for a liver biopsy and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-03-02 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Postprandial phosphoproteomic changes in liver tissue in healthy individuals | 60 minutes after the meal administered at the study day
  Phosphorproteomic changes will be performed using MS-based approach that allows identification of phosphorylations sites at proteins in the liver. The comparison will be done between 'fasted' and 'postprandial' samples

SECONDARY OUTCOMES:
Postprandial phosphoproteomic changes in liver tissue between healthy participants and patients with cirrhosis or patients with NAFLD. | 60 minutes after the meal administered at the study day
  Phosphorproteomic changes will be performed using MS-based approach that allows identification of phosphorylations sites at proteins in the liver. The comparison will be done between 'fasted' and 'postprandial' samples
Postprandial proteomic, metabolomic and transcriptomic changes in liver tissue in healthy individuals and compared to patients with cirrhosis and patients with NAFLD | 60 minutes after the meal administered at the study day
  Proteomic, metabolomic and transcriptomic changes will be performed using MS-based approaches and Next generation sequencing that allows identification of proteins, metabolites, RNA-transcripts in the liver. The comparison will be done between 'fasted' and 'postprandial' samples
Postprandial proteomic, metabolomic and Peptidomic changes in blood obtained from liver vein and peripheral vein in healthy individuals and compared to patients with cirrhosis and patients with NAFLD | 120 minutes after the meal administered at the study day
  Proteomic, metabolomic and hormonal changes will be performed using MS-based approaches and ELISAs that allows identification and measurements of proteins, metabolites and hormones from the liver. The comparison will be done between 'fasted' and 'postprandial' samples
Effect of exogenous glucagon on changes in liver phosphoproteomics, proteomics, metabolomics, and transcriptomics in healthy individuals. | 30 minutes after the meal administered at the study day
  Proteomic, metabolomic and transcriptomic changes will be performed using MS-based approaches and Next generation sequencing that allows identification of proteins, metabolites, RNA-transcripts in the liver. The comparison will be done between 'fasted' and samples obtained after glucagon injection
Effect of exogenous glucagon on changes in phosphoproteomics, proteomics, metabolomics and peptidomic in blood obtained from liver vein and peripheral vein in healthy individuals | 120 minutes after the meal administered at the study day
  Proteomic, metabolomic and hormonal changes will be performed using MS-based approaches and ELISAs that allows identification and measurements of proteins, metabolites and hormones from the liver. The comparison will be done between 'fasted' and samples obtained after glucagon injection

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Jacob Wewer Albrechtsen, MD, Assoc. Prof., Principal Investigator — NNF Center for Protein Research, Faculty of Health and Medical Sciences, University of Copenhagen, Denmark; Lise Lotte Gluud, MD, Prof, Principal Investigator — Gastrounit, Copenhagen University Hospital Hvidovre, Denmark
Locations (1):
- Gastrounit, Copenhagen University Hospital Hvidovre, Hvidovre, Capital Region Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://researchleaderprogramme.com/recipients/nicolai-wewer-albrechtsen/